CLINICAL TRIAL: NCT01116219
Title: Bevacizumab, Pemetrexed and Cisplatin, or Erlotinib and Bevacizumab for Advanced Non-Squamous NSCLC Stratified by EGFR Mutation Status. A Multicenter Phase II Trial Including Biopsy at Progression (BIO-PRO Trial).
Brief Title: Bevacizumab, Pemetrexed Disodium, and Cisplatin or Erlotinib Hydrochloride and Bevacizumab in Treating Patients With Stage IV Non-Small Cell Lung Cancer. A Multicenter Phase II Trial Including Biopsy at Progression (BIO-PRO Trial).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 19/09; SWS-SAKK-19-09; EU-21026
Record Dates: First submitted 2010-04-27; First posted 2010-05-04 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Lung Cancer
Keywords: adenocarcinoma of the lung; bronchoalveolar cell lung cancer; large cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar; Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Erlotinib Hydrochloride; Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stratum mut EGFR (Active Comparator): * Bevacizumab 7.5 mg/kg i.v. every 3 weeks and
  * Erlotinib 150 mg p.o. daily until progression.
  Interventions: Biological: bevacizumab, erlotinib
- Stratum wtEGFR (Active Comparator): Cohort 1:
  Induction chemotherapy with
  * Bevacizumab 7.5 mg/kg i.v. and
  * Pemetrexed 500 mg/m2 i.v. and
  * Cisplatin* 75 mg/m2 i.v. every 3 weeks for a maximum of 4 cycles or until progression.
  Followed by maintenance therapy in patients without disease progression with
  * Bevacizumab 7.5 mg/kg i.v. and
  * Pemetrexed 500 mg/m2 i.v. every 3 weeks until progression.
  Cohort 2:
  Induction chemotherapy with
  * Pemetrexed 500 mg/m2 i.v. and
  * Cisplatin* 75 mg/m2 i.v. every 3 weeks for a maximum of 4 cycles or until progression.
  Followed by maintenance therapy in patients without disease progression with
  o Pemetrexed 500 mg/m2 i.v. every 3 weeks until progression.
  Interventions: Drug: bevacizumab, pemetrexed, cisplatin

INTERVENTIONS:
Biological: bevacizumab, erlotinib — * Bevacizumab 7.5 mg/kg i.v. every 3 weeks and
  * Erlotinib 150 mg p.o. daily until progression.
  Other Names: bevacizumab (Avastin); erlotinib (Tarceva)
  Arms: Stratum mut EGFR
Drug: bevacizumab, pemetrexed, cisplatin — Induction chemotherapy with
  * Bevacizumab 7.5 mg/kg i.v. and
  * Pemetrexed 500 mg/m2 i.v. and
  * Cisplatin* 75 mg/m2 i.v. every 3 weeks for a maximum of 4 cycles or until progression. Followed by maintenance therapy in patients without disease progression with
  * Bevacizumab 7.5 mg/kg i.v. and
  * Pemetrexed 500 mg/m2 i.v. every 3 weeks until progression.
  Other Names: Bevacizumab (Avastin); pemetrexed (Alimta)
  Arms: Stratum wtEGFR

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as pemetrexed disodium and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether bevacizumab given together with pemetrexed disodium and cisplatin is more effective than erlotinib hydrochloride given together with bevacizumab in treating patients with non-small cell lung cancer.

PURPOSE: This phase II trial is studying giving bevacizumab together with pemetrexed disodium and cisplatin to see how well it works compared with giving erlotinib hydrochloride together with bevacizumab in treating patients with stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To demonstrate that tailored therapy, according to tumor histology and EGFR-mutation status, and the introduction of novel drug combinations in the frontline treatment of patients with stage IV non-squamous non-small cell lung cancer, is promising for further investigation.

Secondary

* To prospectively explore molecular markers of clinical outcomes.

OUTLINE: This is a multicenter study. Patients are stratified according to EGFR(epidermal growth factor receptor)-mutation status (mutated vs wildtype). Patients are assigned to 1 of 2 groups.

* mutEGFR (mutated epidermal growth factor receptor) group: Patients receive bevacizumab IV over 30-90 minutes on day 1 and oral erlotinib hydrochloride once daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
* wtEGFR (wildtype epidermal growth factor receptor) group cohort 1:

  * Induction chemotherapy: Patients receive bevacizumab IV over 30-90 minutes, pemetrexed disodium IV over 10 minutes, and cisplatin IV over 60 minutes on day 1. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  * Maintenance therapy: Patients without progressive disease receive bevacizumab IV over 30-90 minutes and pemetrexed disodium IV over 10 minutes on day 1. Treatment repeats every 21 days in the absence of disease progression.

Blood and tissue specimens are collected for EGFR and molecular markers analysis, including gene expression, mutation, and pharmacogenomic analyses.

After completion of study treatment, patients are followed every 3 months.

* wtEGFR (wildtype epidermal growth factor receptor) group cohort 2:

  * Induction chemotherapy: Patients receive pemetrexed disodium IV over 10 minutes, and cisplatin IV over 60 minutes on day 1. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  * Maintenance therapy: Patients without progressive disease receive pemetrexed disodium IV over 10 minutes on day 1. Treatment repeats every 21 days in the absence of disease progression.

Blood and tissue specimens are collected for EGFR and molecular markers analysis, including gene expression, mutation, and pharmacogenomic analyses.

After completion of study treatment, patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 129 evaluable patients (77 in cohort 1 and 52 in cohort 2) with wtEGFR status and 20 patients with mutEGFR status will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell lung cancer of the following non-squamous subtypes:

  * Adenocarcinoma
  * Bronchioloalveolar carcinoma
  * Large cell carcinoma
* Stage IV disease including any of the following:

  * M1a (separate tumor nodule in a contralateral lobe, tumor with pleural nodules, or malignant pleural or pericardial effusion)
  * M1b (distant metastasis)
* Measurable disease, defined as ≥ 1 lesion (outside of irradiated areas) that can be measured in ≥ 1 dimension as ≥ 10 mm (≥ 15 mm in case of lymph nodes) according to RECIST 1.1
* Paraffin-embedded or formalin-fixed diagnostic biopsy collected in the past 2 months must be available
* Must have EGFR-mutation status (mutated or wild type) confirmed by the central pathologist in Basel
* Must consent to tumor biopsy at progression
* No intrathoracic tumors invading or abutting major blood vessels
* No CNS metastases by mandatory CT scan (MRI within the past 3 weeks is acceptable)

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Hemoglobin ≥ 100 g/L
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT ≤ 3 times ULN (≤ 5 times ULN if liver metastases are present)
* Alkaline phosphatase ≤ 3 times ULN (≤ 5 times ULN if liver metastases are present)
* Calculated creatinine clearance ≥ 60 mL/min
* Urine dipstick for proteinuria < 2+
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 months after completion of study therapy
* Must be compliant and have geographic proximity to allow proper staging and follow-up
* No active bleeding, including hemoptysis ≥ grade 2 (defined as bright red blood of ≥ 5 mL per episode within the past 4 weeks)

  * Minor hemoptysis is allowed
* No prior malignancy within the past 5 years, except adequately treated cervical carcinoma in situ or localized non-melanoma skin cancer
* No psychiatric disorder precluding understanding of information on trial-related topics, giving informed consent, or interfering with compliance for oral drug intake
* No other medical condition that would impair the ability of the patient to participate in the trial or might preclude therapy with trial drugs, including any of the following:

  * Unstable or uncompensated respiratory, cardiac, hepatic, or renal disease
  * Active infection
  * Uncontrolled diabetes mellitus
  * Uncontrolled arterial hypertension (i.e., BP ≥ 150/100 mm Hg despite optimal medical therapy)
  * History of myocardial infarction in the last 3 months
  * History of hemorrhagic disorders
  * Non-healing wound, ulcer, or bone fracture
  * Significant traumatic injury within the past 28 days
* No known hypersensitivity to trial drugs or to any other component of the trial drugs

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy or molecular-targeted therapy for metastatic disease (neoadjuvant or adjuvant chemotherapy allowed if terminated > 6 months ago)
* No prior radiotherapy to lesion(s) selected for measurement
* At least 30 days since prior yellow fever vaccination
* At least 30 days since prior experimental drugs, anticancer therapy, or treatment in a clinical trial
* More than 28 days since major surgical procedure or open biopsy
* No concurrent full-dose oral, intravenous, or subcutaneous anticoagulants (low-dose heparin or aspirin [≤ 325 mg p.o. daily] allowed)
* No concurrent herbal extracts or drugs contraindicated for use with trial drugs
* No concurrent investigational agents
* No other concurrent anti-neoplastic or anti-tumor agents, including chemotherapy, immunotherapy, or hormonal anticancer therapy
* No concurrent Asasantin® (acetylsalicylic acid and dipyridamole) or Plavix® (clopidogrel bisulfate)

Inclusion criteria

* Before registration, patient must give written informed consent for participation in the trial including tumor biopsy at progression.
* Patient must have the capability to understand informed consent and information given by the investigator on the trial.
* Non-small cell lung cancer (NSCLC), predominant non-squamous subtype (adenocarcinoma, bronchioloalveolar carcinoma, and large cell carcinoma) confirmed by the central pathologist in Basel.
* NSCLC stage IV according to the 7th edition of the TNM classification, including M1a (separate tumor nodule in a contralateral lobe, tumor with pleural nodules or malignant pleural or pericardial effusion) and/or M1b (distant metastasis).
* Most recent diagnostic biopsy paraffin-embedded or only formalin-fixed and sufficient for further molecular analysis as determined by central pathologist in Basel.
* EGFR mutation status determined by local or central pathologist in Basel.
* EDTA blood samples (2 x 5 mL) for translational research projects will be taken before treatment start.
* WHO performance status 0-1 (see Appendix 4).
* Age ≥ 18 years and legally competent person.
* Measurable disease, defined as at least one lesion (outside of irradiated areas) that can be measured in at least one dimension as ≥ 10 mm (≥ 15 mm in case of lymph nodes)according to RECIST v1.1
* Adequate hematological values: Hemoglobin ≥ 100 g/L, neutrophils ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L
* Adequate hepatic function: Bilirubin ≤ 1.5 x ULN, ALT and AP ≤ 3 x ULN (≤ 5 x ULN in case of liver metastases)
* Adequate renal function: Calculated creatinine clearance ≥ 60 mL/min (according to the formula of Cockroft-Gault)
* Urine dipstick for proteinuria < 2+
* Women are not breastfeeding. Women with child-bearing potential are using effective contraception (see 9.2.4 and 9.3.5), are not pregnant and agree not to become pregnant during participation in the trial and during the 12 months thereafter. A negative pregnancy test before inclusion into the trial is required for all women with childbearing potential. Men agree not to father a child during participation in the trial or during the 12 months thereafter.
* Patient compliance and geographic proximity allow proper staging and follow-up.

Exclusion criteria

* Diagnosis of SCLC, predominantly squamous NSCLC (>50% by central pathology review) or combined SCLC-NSCLC.
* Patients with intrathoracic tumors invading or abutting major blood vessels.
* Prior chemotherapy or molecular targeted therapy for metastatic disease, with the exception of neoadjuvant or adjuvant chemotherapy if terminated 6 months before registration. Prior radiotherapy to lesion(s) selected for measurement.
* CNS metastases by mandatory CT-scan (MRI is acceptable).
* Anticoagulation, with the exception of low dose heparin or aspirin (≤ 325 mg p.o. daily).
* Active bleeding, including hemoptysis ≥ grade 2 (defined as bright red blood of at least 5 mL per episode within the last 4 weeks of registration). Minor hemoptysis is allowed.
* Yellow fever vaccination within the 30 days prior to registration.
* Previous malignancy within 5 years with the exception of adequately treated cervical carcinoma in situ or localized non-melanoma skin cancer.
* Psychiatric disorder precluding understanding of information on trial related topics, giving informed consent, or interfering with compliance for oral drug intake.
* Concurrent treatment with other experimental drugs or other anti-cancer therapy, treatment in a clinical trial within 30 days prior to trial entry.
* Evidence of other medical condition which would impair the ability of the patient to participate in the trial or might preclude therapy with trial drugs (e.g. unstable or uncompensated respiratory, cardiac, hepatic or renal disease, active infection, uncontrolled diabetes mellitus; uncontrolled arterial hypertension ≥ 150/100 mmHg, history of myocardial infarction in the last 3 months, history of hemorrhagic disorders, non healing wound, ulcer or bone fracture)
* Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to registration
* Known hypersensitivity to trial drugs or hypersensitivity to any other component of the trial drugs.
* Any concomitant drugs contraindicated for use with the trial drugs according to the Swissmedic-approved product information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Estimated)
Dates: Start 2010-06; Primary Completion 2014-07 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Progression-free survival at 6 months in stratum wtEGFR cohort 1 | at 6 months

SECONDARY OUTCOMES:
Progression-free survival | at 6 months
Overall survival | from registration until death
Best response (RECIST 1.1) | up to disease progression or start of new treatment
Adverse events (CTCAE v4.0)
Molecular markers in tumor tissue and blood

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Gautschi, MD, Study Chair — Luzerner Kantonsspital; Adrian Ochsenbein, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern; Nicolas Mach, MD, Principal Investigator — Hopital Cantonal Universitaire de Geneve HUG; Sacha Rothschild, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (22):
- Switzerland (22):
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Saint Claraspital AG, Basel
  - Clinical Cancer Research Center at University Hospital Basel, Basel
  - Istituto Oncologico della Svizzera Italiana - Ospedale San Giovanni, Bellinzona
  - Inselspital Bern, Bern
  - Spitalzentrum Biel, Biel
  - Kantonsspital Bruderholz, Bruderholz
  - Kantonsspital Graubuenden, Chur
  - Kantonsspital Freiburg, Fribourg
  - Hopital Cantonal Universitaire de Geneve, Geneva
  - Centre Pluridisciplinaire d' Oncologie, Lausanne
  - Kantonsspital Liestal, Liestal
  - Kantonsspital Luzern, Luzerne
  - Kantonsspital Olten, Olten
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Regionalspital, Thun
  - Spital Uster, Uster
  - Kantonsspital Winterthur, Winterthur
  - Onkozentrum Hirslanden, Zurich
  - UniversitaetsSpital Zuerich, Zurich
  - City Hospital Triemli, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gautschi O, Rothschild SI, Li Q, Matter-Walstra K, Zippelius A, Betticher DC, Fruh M, Stahel RA, Cathomas R, Rauch D, Pless M, Peters S, Froesch P, Zander T, Schneider M, Biaggi C, Mach N, Ochsenbein AF; Swiss Group for Clinical Cancer Research. Bevacizumab Plus Pemetrexed Versus Pemetrexed Alone as Maintenance Therapy for Patients With Advanced Nonsquamous Non-Small-cell Lung Cancer: Update From the Swiss Group for Clinical Cancer Research (SAKK) 19/09 Trial. Clin Lung Cancer. 2017 May;18(3):303-309. doi: 10.1016/j.cllc.2016.11.007. Epub 2016 Nov 23. PMID 27993482